CLINICAL TRIAL: NCT03075748
Title: Visceral Manifold Study for the Repair of Thoracoabdominal Aortic Aneurysms
Brief Title: Visceral Manifold Study for the Repair of TAAA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Medtronic (Industry); Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-01-001 Visceral Manifold
Record Dates: First submitted 2017-02-24; First posted 2017-03-09 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Thoracoabdominal Aortic Aneurysms
Keywords: Vascular; Stent; Graft
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Primary study (Experimental): Patients meeting primary inclusion/exclusion criteria will be enrolled in primary study arm and be treated with the TAAA Debranching Stent Graft System.
  Interventions: Device: TAAA Debranching Stent Graft System
- Expanded selection (Experimental): Patients who fail to meet inclusion criteria for the primary study arm may be enrolled under the expanded selection arm and be treated with the TAAA Debranching Stent Graft System.
  Interventions: Device: TAAA Debranching Stent Graft System

INTERVENTIONS:
Device: TAAA Debranching Stent Graft System — The TAAA Debranching Stent Graft System is made up of two main body components and makes use of several off-the-shelf FDA-approved stent graft components. The two custom main body grafts are the thoracic bifurcation and the visceral manifold. The thoracic bifurcation is deployed in the thoracic aorta and provides the proximal seal for the device. The two limbs of the thoracic bifurcation allows for continued aortic flow while deploying the visceral segment. The visceral manifold is deployed within the larger 20 mm limb of the thoracic bifurcation to set the stage for the visceral debranching. The branches of the visceral manifold extend to the visceral vessel with the use of covered bridging stents and provide distal seal of the manifold.

SUMMARY:
The outcomes from prior clinical evaluation of the study device, including successfully treating 99% (84/85) of the intended target vessels and 96% (27/28) limb patency observed at one year, demonstrate the potential benefits of the device. When contrasted with open repair's significant complication rates and branch fenestrated device's significant anatomic and logistic limitations, the potential risk of the proposed novel graft does not outweigh the potential benefit of widened anatomic availability and improved patency rates. Given the potential benefits, the investigators feel that it is justified to expose the target patient population to the potential risk. The non-clinical testing performed by Medtronic and the clinical results reported by Sanford Health show adequate safety of the device to support an early feasibility study.

The investigators would like to perform an early feasibility study under a defined and controlled protocol to collect prospective preliminary safety and device functionality data. The investigators believe an early feasibility study is most appropriate for this novel approach. The limited sample size allows adequate patient data to be collected under a controlled protocol without exposing a large patient population to the risk associated with a novel device design.

DETAILED DESCRIPTION:
This study is a prospective, single-center, non-randomized, single-arm study to evaluate the therapeutic benefit of the TAAA Debranching Stent Graft System. A total of 15 patients will be enrolled in the study.

* 10 subjects total will be treated in the primary study arm
* 5 subjects total will be treated in the expanded selection arm

The duration of the Investigation is anticipated as follows:

* Time to Complete Enrollment: 24 months
* Subject Follow-up Time: 5 years from last subject enrollment
* Total Duration Time: 7 years

The primary objective of the clinical investigation "Visceral Manifold Study for the repair of thoracoabdominal aortic aneurysms" is to assess the use of the TAAA Debranching Stent Graft System to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy. The primary intent of the study is to assess safety acutely (i.e. freedom from major adverse events (MAE) at 30 days) and preliminary effectiveness (i.e., treatment success and technical success) of the device acutely (i.e., the proportion of treatment group subjects that achieve and maintain treatment success at one year).

Additionally, the study will assess technical success and treatment success at each follow-up interval.

ELIGIBILITY:
Primary Study Arm

Inclusion Criteria:

* A patient may be entered into the study if the patient has at least one of the following:

  * An aneurysm with a maximum diameter of > 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
  * Aneurysm with a history of growth > 0.5 cm in 6 months
  * Saccular aneurysm deemed at significant risk for rupture
  * Symptomatic aneurysm greater than 4.5 cm
* Axillary or brachial and iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
* Proximal landing zone for the thoracic bifurcation stent graft that has:

  * ≥ 2.5 cm of nonaneurysmal aortic segment including previously placed graft material (neck) distal to the left subclavian artery (LSA) diameter in the range of 26-42 mm
  * Adequate distance from the celiac artery, in order to accommodate cannulation from the antegrade access point when considering the total deployed length of the thoracic bifurcation and visceral manifold
* Minimum branch vessel diameter greater than 5 mm
* Iliac artery or aortic distal fixation site, including both native tissue and previously placed graft, greater than or equal to 15 mm in length and diameter in the range of 8 - 25 mm
* Age: ≥ 18 years old
* Life expectancy: > 1 year

Exclusion Criteria:

General exclusion

* Patient is a good candidate for and elects for open surgical repair
* Can be treated in accordance with the instructions for use with a legally marketed endovascular prosthesis
* Is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Urgent or emergent presentation
* Patient is pregnant or breastfeeding
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a dissection in the portion of the aorta intended to be treated
* Obstructive stenting of any or all of the visceral vessels
* Poor performance status including two major system failures (cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)

Medical exclusion criteria

* Known sensitivities or allergies to the materials of construction of the devices, including nitinol (Nickel: Titanium), polyester, platinum-iridium, polytetrafluoroethylene (PTFE), platinum, gold, polyethylene, or stainless steel.
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
* Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection
* Baseline creatinine greater than 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome)

Anatomical exclusion criteria

* Thrombus or excessive calcification within the neck of the aneurysm
* Anatomy that would not allow maintenance of at least one patent hypogastric artery
* Anatomy that would not allow primary or assisted patency of the left subclavian artery

Expanded Selection Criteria Subjects who fail to meet inclusion criteria for the primary study arm may be enrolled under an expanded selection arm if they meet the following criteria.

Inclusion Criteria

* Patient that meets the criteria for inclusion in the primary study arm but has one or more of the following criteria which would exclude them from the primary study arm:

  * Minimum branch vessel diameter less than 5 mm
  * Urgent or emergent presentation
  * Patient has a contained rupture
  * Patient has a ruptured aneurysm
  * Patient has a type B dissection (subacute or chronic) in the portion of the aorta intended to be treated
  * Poor performance status including two major system failures (cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)
  * Baseline creatinine greater than 2.0 mg/dL
  * Anatomy that would not allow for maintenance of at least one hypogastric artery
  * Anatomy that would not allow for primary or assisted patency of the left subclavian artery Or
* Patient that meets the criteria for inclusion in the primary study arm and:

  * Would not be eligible for the primary study arm per a documented reason other than those outlined above, and
  * Per the opinion of the Principal Investigator, with concurrence of the IRB, alternative therapies are unsatisfactory and the probable risk of using the investigational device is no greater than the probable risk from the disease or condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects free from major adverse events | 30 days
  Primary safety outcome: Major adverse events include death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and stroke
Proportion of subjects with treatment success | at 1 year
  Primary effectiveness outcome: Treatment success is defined as a composite of technical success and freedom from the following: aneurysm enlargement, aneurysm rupture, aneurysm-related mortality, conversion to open repair, secondary intervention for migration, Type I and III endoleaks, device integrity failure, and patency-related events

SECONDARY OUTCOMES:
Proportion of subjects with technical success | 5 years
Proportion of subjects free from individual components of primary safety endpoint | at 30 days
  Individual components of primary safety endpoint include: death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, stroke
Proportion of subjects free from paraparesis | 30 days
  Free from paraparesis
Proportion of subjects with treatment success | 5 years
  Treatment success includes freedom from: aneurysm enlargement; aneurysm-related mortality; aneurysm rupture; conversion to open repair; secondary intervention for migration, type I and III endoleaks, device integrity failure (i.e. fracture), and patency-related events (i.e. device stenosis or occlusion and embolic events); renal failure; all-cause mortality; endoleaks; device integrity failure (e.g. fracture); patency-related events (i.e. device stenosis or occlusion and embolic events); other device-related events

CONTACTS AND LOCATIONS:
Overall Officials: Murray Shames, MD, Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - Tampa General Hospital/ University of South Florida, Tampa, Florida
  - University of South Florida - South Tampa Campus, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with Sanford Health

REFERENCES:
- [Result] Anderson J, Nykamp M, Danielson L, Remund T, Kelly PW. A novel endovascular debranching technique using physician-assembled endografts for repair of thoracoabdominal aneurysms. J Vasc Surg. 2014 Nov;60(5):1177-1184. doi: 10.1016/j.jvs.2014.05.090. Epub 2014 Jul 3. PMID 24997805
- [Result] Anderson J, Nykamp M, Remund T, Kelly P. Complete endovascular debranching of the aortic arch: A report of two cases. Vascular. 2015 Jun;23(3):310-5. doi: 10.1177/1708538114542174. Epub 2014 Jul 11. PMID 25015113
- [Result] Danielson L, Anderson J, Nykamp M, Remund T, Kelly P. Treatment of a massive left femoral arteriovenous malformation using an innovative modular hybrid bifurcated stent graft system. Ann Vasc Surg. 2014 May;28(4):1031.e15-20. doi: 10.1016/j.avsg.2013.07.023. Epub 2013 Oct 31. PMID 24184461
- [Result] Narayanan S, Shalhoub J, Karunanithy N, Burfitt N. Primary suture-anastomosis of the Viabahn endoprosthesis to a native artery. J Vasc Surg. 2010 May;51(5):1297-9. doi: 10.1016/j.jvs.2009.12.045. Epub 2010 Mar 19. PMID 20303692
- [Result] Donas KP, Lachat M, Rancic Z, Oberkofler C, Pfammatter T, Guber I, Veith FJ, Mayer D. Early and midterm outcome of a novel technique to simplify the hybrid procedures in the treatment of thoracoabdominal and pararenal aortic aneurysms. J Vasc Surg. 2009 Dec;50(6):1280-4. doi: 10.1016/j.jvs.2009.06.053. PMID 19958984
- [Result] Oderich GS, Fatima J, Gloviczki P. Stent graft modification with mini-cuff reinforced fenestrations for urgent repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2011 Nov;54(5):1522-6. doi: 10.1016/j.jvs.2011.06.023. Epub 2011 Sep 16. PMID 21925826